CLINICAL TRIAL: NCT00021866
Title: Neurodevelopmental Effects of Antiepileptic Drugs II: the NEAD Study
Brief Title: Developmental Effects On Children Of Women Who Take Antiepileptic Drugs During Pregnancy
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Kimford J. Meador, MD, Professor, Emory University
Other Study IDs: 0334-2001; 2R01NS038455 (NIH); 2R01NS038455-06 (NIH)
Record Dates: First submitted 2001-08-08; First posted 2001-08-10 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-09

CONDITIONS: Epilepsy; Seizure; Cognition Disorders
Keywords: epilepsy; seizure; pregnancy; antiepileptic; AED; carbamazepine; phenytoin; valproate; lamotrigine; child; behavior
MeSH Terms: conditions — Epilepsy; Seizures; Cognition Disorders; Behavior | interventions — amsonic acid; Neuropsychological Tests; Psychological Tests

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood for AED levels Cord Blood for G6PD, Homocysteine Saliva for drug metabolizing enzymes, antioxidant enzymes, DNA repair enzymes, drug membrane transporter proteins and folate-related genes
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Carbamazepine: Children and their mothers exposed to Carbamazepine monotherapy in utero
  Interventions: Behavioral: Differential Abilities Scale; Behavioral: Neuropsychological Testing
- Phenytoin: Children and their mothers exposed to phenytoin in utero
  Interventions: Behavioral: Differential Abilities Scale; Behavioral: Neuropsychological Testing
- Lamotrigine: Children and their mothers exposed to Lamotrigine in utero
  Interventions: Behavioral: Differential Abilities Scale; Behavioral: Neuropsychological Testing
- Valproate: Children and their mothers exposed to Valproate in utero
  Interventions: Behavioral: Differential Abilities Scale; Behavioral: Neuropsychological Testing

INTERVENTIONS:
Behavioral: Differential Abilities Scale — IQ measurement at 3, 4.5 and 6 years of age
  Other Names: DAS
Behavioral: Neuropsychological Testing — Tests of memory, attention, and behavior administered at 2,3, 4.5 and 6 Years of age
  Other Names: (Toni-3) Test of Nonverbal Intelligence; (WAIS) - Wechslers Adult Intelligence Scale -revised; Beck Depression Inventory; Bayley Scales of Infant Development,; NEPSY; Trails Preschool; Preschool Language Scale-4; Expressive One-Word Vocabulary TEst; Peabody Picture Vocabulary Test; Developmental Test of Visual-Motor Integration; Children's Memory Scale; Grooved Pegboard; Bracken Basic Concepts Scale; Wide Range Achievement TEst; Adaptive Behavior Assessment Scale; Behavioral Assessment for Children; Parenting Stress Index

SUMMARY:
The purpose of this study is to determine if antiepileptic drugs (AEDs) differ in their neurodevelopmental effects. Specifically, do the children of the women with epilepsy differ in their behavioral and cognitive development depending on which AED their mother takes during pregnancy?

DETAILED DESCRIPTION:
This is a prospective investigation enrolling 285 to 380 women with epilepsy during the first two trimesters of their pregnancies. There are 25 clinical centers as well as the database center. The women will be taking one of the following AEDs: carbamazepine, phenytoin, valproate, or lamotrigine. Cognitive and behavioral testing of the child will be done up to the age of 6 years. The study does not change the woman's doctor and does not interfere with the care of the treating physician.

ELIGIBILITY:
* Subject must be diagnosed with partial seizures and/or secondary generalization or primary generalized seizures (absence, atonic, myoclonic, and generalized tonic-clonic seizures)
* Subjects must be on either carbamazepine, lamotrigine, phenytoin, or valproate monotherapy.
* Mothers must not have a history of drug abuse (including alcohol) in the last year and have no sequelae of drug abuse.
* Mothers must be able to maintain an accurate seizure diary of major motor seizures
* Subjects must have an IQ greater than or equal to 70 points.
* Subjects must have a history of a negative RPR and HIV.
* Subjects must not have progressive cerebral disease or presence of other major medical illness
* Subjects must not have exposure to known teratogens during pregnancy, except AEDs.
* Subjects must not have poor compliance with prenatal care.
* Subjects must have adequate reading skills to perform the cognitive tests.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mothers and their child(ren) who were exposed to one of the following monotherapies in utero- Lamotrigine, Carbamazepine, Phenytoin, or Valproate. Fathers of the children and a first degree materal relative of the mother are also invited to have IQ testing and medical history
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2000-09; Primary Completion 2010-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Child IQ as measured by the Differential Abilities Scale at 6 Years of age | 6 years

SECONDARY OUTCOMES:
Executive Functioning,Tower-NEPSY | 6 Years
Linguistic Functioning via Expressive one word vocabulary test and NEPSY subscales | 6 Years
Visual-Spatial Motor Functioning via NEPSY subscale and Visual-Motor Integration Scale | 6 Years
Memory via Children's Memory Scale | 6 Years
Motor Functioning via Grooved Pegboard | 6 Years
Academic Functioning via Wide Range Achievement Test | 6 Years
Adaptive Functioning via Adaptive Behavior System -2nd Edition | 6 Years
Behavior via Behavior Assessment for Children & Parent Stress Index | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Kimford J. Meador, M.D., Principal Investigator — Emory University, Atlanta
Locations (21):
- United States (20):
  - University of Alabama, Birmingham, Alabama
  - Arizona Health Sciences, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - RUSH University Medical Center, Chicago, Illinois
  - Via Christi Medical Center, Wichita, Kansas
  - Brigham & Womens' Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Epilepsy Group, Saint Paul, Minnesota
  - Columbia University, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Riddle Health Care II, Media, Pennsylvania
  - Baylor Medical Center, Irving, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- University of Liverpool, Liverpool, United Kingdom

REFERENCES:
- [Result] Meador KJ, Chadwick D, Clayton-Smith J, Pennell P, Liporace J, Kalayian L, and NEAD Study Group. Antiepileptic drugs in pregnancy: Differences in U.K. and U.S.A. Epilepsia, 2003;44 (Suppl. 9):289.
- [Result] Meador KJ, Page P, Liporace J, Kalayjian L, NEAD Study Group. Antiepileptic Drugs in Pregnancy. Neurology 2004;62 (Suppl 5):A311.
- [Result] Meador KJ, Baker GA, Clayton Smith J, Pennell P, Liporace J, Kalayjian L, Kini U, NEAD Study Group. Differential Effects of Antiepileptic Drugs on Serious Adverse Outcomes in Children Exposed In Utero. Epilepsia 2004;45 (Suppl 3):58
- [Result] Meador KM, Loring DW, Baker G, Smith JC, Pennell P, Liporace J, Kalayjian L, Kini U, NEAD Study Group. Differential and dose dependent effects of in utero antiepileptic drugs. Neurology 2005;64 (Suppl 1):A427
- [Result] Meador KJ, Baker GA, Finnell RH, Kalayjian LA, Liporace JD, Loring DW, Mawer G, Pennell PB, Smith JC, Wolff MC; NEAD Study Group. In utero antiepileptic drug exposure: fetal death and malformations. Neurology. 2006 Aug 8;67(3):407-12. doi: 10.1212/01.wnl.0000227919.81208.b2. PMID 16894099
- [Derived] Meador KJ, Pennell PB, May RC, Brown CA, Baker G, Bromley R, Loring DW, Cohen MJ; NEAD Investigator Group. Effects of periconceptional folate on cognition in children of women with epilepsy: NEAD study. Neurology. 2020 Feb 18;94(7):e729-e740. doi: 10.1212/WNL.0000000000008757. Epub 2019 Dec 23. PMID 31871217
- [Derived] Meador KJ, Baker GA, Browning N, Cohen MJ, Bromley RL, Clayton-Smith J, Kalayjian LA, Kanner A, Liporace JD, Pennell PB, Privitera M, Loring DW; Neurodevelopmental Effects of Antiepileptic Drugs (NEAD) Study Group. Breastfeeding in children of women taking antiepileptic drugs: cognitive outcomes at age 6 years. JAMA Pediatr. 2014 Aug;168(8):729-36. doi: 10.1001/jamapediatrics.2014.118. PMID 24934501
- [Derived] Meador KJ, Baker GA, Browning N, Cohen MJ, Bromley RL, Clayton-Smith J, Kalayjian LA, Kanner A, Liporace JD, Pennell PB, Privitera M, Loring DW; NEAD Study Group. Fetal antiepileptic drug exposure and cognitive outcomes at age 6 years (NEAD study): a prospective observational study. Lancet Neurol. 2013 Mar;12(3):244-52. doi: 10.1016/S1474-4422(12)70323-X. Epub 2013 Jan 23. PMID 23352199
- See also: Click here for more information about this study and a list of recruiting centers — https://web.emmes.com/study/monead